CLINICAL TRIAL: NCT00049309
Title: Prostate Cancer: Impact Of Fat And Flaxseed - Modified Diets
Brief Title: Low-Fat Diet and/or Flaxseed in Preventing Prostate Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pro00008602; DUMC-1385-02-7R3ER; NCI-P02-0235; CCUM-0202; UMCC-0202; CDR0000258042 (Other: NCI)
Record Dates: First submitted 2002-11-12; First posted 2003-01-27 (Estimated); Last update posted 2017-02-23 (Actual); Status verified 2013-02

CONDITIONS: Prostate Cancer
Keywords: stage I prostate cancer; stage IIB prostate cancer; stage IIA prostate cancer; stage III prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Diet Therapy; Linseed Oil

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Control (No Intervention): Usual diet
- Flaxseed diet (Experimental): 30 gram flaxseed dietary modification
  Interventions: Dietary Supplement: flaxseed
- Low fat diet (Experimental): Low fat dietary modification
  Interventions: Dietary Supplement: dietary intervention
- Low fat + Flaxseed diet (Experimental): Low fat and 30 gram flaxseed dietary modification
  Interventions: Dietary Supplement: dietary intervention; Dietary Supplement: flaxseed

INTERVENTIONS:
Dietary Supplement: dietary intervention
  Arms: Low fat + Flaxseed diet; Low fat diet
Dietary Supplement: flaxseed
  Arms: Flaxseed diet; Low fat + Flaxseed diet

SUMMARY:
RATIONALE: A diet that is low in fat and/or high in flaxseed may slow or prevent disease progression of prostate cancer.

PURPOSE: Randomized phase II trial to study the effectiveness of a diet that is low in fat and/or high in flaxseed in slowing or preventing disease progression in patients who have newly diagnosed prostate cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare tumor proliferation in patients with newly diagnosed prostate cancer eating fat- and/or flaxseed-modified diets.
* Compare differences in histopathological markers associated with prostate cancer (rates of apoptosis, extent of high-grade prostatic intraepithelial neoplasia) among patients in these diet groups.
* Compare changes in serum prostate specific antigen among patients in these diet groups.
* Compare changes in hormone-related factors (total serum testosterone and free androgen index, insulin-like growth factor [IGF], and IGF-binding protein-3) among patients in these diet groups.
* Compare the effects of diet on nutritional biomarkers (levels of lignans in the urine and ejaculate, fatty acid profiles of erythrocytes and prostatic tissue) in these patients.
* Determine associations between dietary modification and changes in dietary biomarkers, hormonal intermediates, and study endpoints in these patients.

OUTLINE: This is a randomized study. Patients are stratified according to Gleason score (less than 7 vs at least 7) and race (black vs non-black). Patients are randomized to 1 of 4 diet groups.

* Arm I (Flaxseed-supplemented diet): Patients are instructed to incorporate ground flaxseed into their daily diets.
* Arm II (Low-fat diet): Patients are instructed on ways to achieve a diet with no greater than 20% of total energy from dietary fat.
* Arm III (Flaxseed-supplemented, low-fat diet): Patients are instructed as in arm I and arm II.
* Arm IV (Control diet): Patients are contacted weekly, but do not receive dietary counseling until after surgery.

All patients ingest the diets for at least 3 weeks and complete diet diaries until surgery. After surgery, all patients receive dietary counseling.

PROJECTED ACCRUAL: A total of 160 patients (40 per treatment arm) will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed prostate cancer
* At least 3 weeks until planned prostatectomy (24 days between day 1 visit and surgery)
* Current diet that provides more than 30% of calories from fat

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* Not specified

Life expectancy

* Not specified

Hematopoietic

* Not specified

Hepatic

* Not specified

Renal

* Not specified

Other

* Mentally competent
* Able to speak and write English
* Must have telephone access

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* Not specified

Endocrine therapy

* No concurrent hormonal therapy

Radiotherapy

* Not specified

Surgery

* At least 2 weeks since prior prostate biopsy

Other

* At least 7 days since prior antibiotics
* No prior therapy for prostate cancer
* No concurrent dietary supplements initiated within the past 3 months or anticipated to begin during study except standard multivitamin/mineral preparations (e.g., One-A-Day, Theragran, or Centrum) that do not supply > 100% of the recommended daily allowance of any vitamin or mineral
* No other concurrent neoadjuvant therapies
* No other concurrent flaxseed consumption

Ages: 18 Years to 120 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 161 (Actual)
Dates: Start 2003-01; Primary Completion 2006-05 (Actual); Study Completion 2006-05 (Actual)

PRIMARY OUTCOMES:
Prostatic Carcinoma Proliferation Rate by MIB-1 assay at time of prostatectomy

SECONDARY OUTCOMES:
Prostatic Carcinoma Apoptotic Index by TUNEL assay at time of prostatectomy
Prostate-specific antigen by Hybritech assay at baseline and follow-up
Total testosterone, sex hormone binding globulin, insulin-like growth factor (IGF), and IGF-binding protein-3, total cholesterol, and low-density lipoprotein cholesterol by ELISA assays at baseline and follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Wendy Demark-Wahnefried, PhD, Study Chair — Duke Cancer Institute
Locations (3):
- United States (3):
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Lineberger Comprehensive Cancer Center at University of North Carolina - Chapel Hill, Chapel Hill, North Carolina
  - Duke Comprehensive Cancer Center, Durham, North Carolina

REFERENCES:
- [Background] Demark-Wahnefried W, Robertson CN, Walther PJ, Polascik TJ, Paulson DF, Vollmer RT. Pilot study to explore effects of low-fat, flaxseed-supplemented diet on proliferation of benign prostatic epithelium and prostate-specific antigen. Urology. 2004 May;63(5):900-4. doi: 10.1016/j.urology.2003.12.010. PMID 15134976
- [Background] Lin X, Gingrich JR, Bao W, Li J, Haroon ZA, Demark-Wahnefried W. Effect of flaxseed supplementation on prostatic carcinoma in transgenic mice. Urology. 2002 Nov;60(5):919-24. doi: 10.1016/s0090-4295(02)01863-0. PMID 12429338
- [Result] Demark-Wahnefried W, Polascik TJ, George SL, Switzer BR, Madden JF, Ruffin MT 4th, Snyder DC, Owzar K, Hars V, Albala DM, Walther PJ, Robertson CN, Moul JW, Dunn BK, Brenner D, Minasian L, Stella P, Vollmer RT. Flaxseed supplementation (not dietary fat restriction) reduces prostate cancer proliferation rates in men presurgery. Cancer Epidemiol Biomarkers Prev. 2008 Dec;17(12):3577-87. doi: 10.1158/1055-9965.EPI-08-0008. PMID 19064574
- [Result] Demark-Wahnefried W, George SL, Switzer BR, Snyder DC, Madden JF, Polascik TJ, Ruffin MT 4th, Vollmer RT. Overcoming challenges in designing and implementing a phase II randomized controlled trial using a presurgical model to test a dietary intervention in prostate cancer. Clin Trials. 2008;5(3):262-72. doi: 10.1177/1740774508091676. PMID 18559416
- [Result] Heymach JV, Shackleford TJ, Tran HT, Yoo SY, Do KA, Wergin M, Saintigny P, Vollmer RT, Polascik TJ, Snyder DC, Ruffin MT 4th, Yan S, Dewhirst M, Kunnumakkara AB, Aggarwal BB, Demark-Wahnefried W. Effect of low-fat diets on plasma levels of NF-kappaB-regulated inflammatory cytokines and angiogenic factors in men with prostate cancer. Cancer Prev Res (Phila). 2011 Oct;4(10):1590-8. doi: 10.1158/1940-6207.CAPR-10-0136. Epub 2011 Jul 15. PMID 21764858
- [Result] Azrad M, Zhang K, Vollmer RT, Madden J, Polascik TJ, Snyder DC, Ruffin MT, Moul JW, Brenner D, Hardy RW, Demark-Wahnefried W. Prostatic alpha-linolenic acid (ALA) is positively associated with aggressive prostate cancer: a relationship which may depend on genetic variation in ALA metabolism. PLoS One. 2012;7(12):e53104. doi: 10.1371/journal.pone.0053104. Epub 2012 Dec 28. PMID 23285256
- [Result] Azrad M, Vollmer RT, Madden J, Dewhirst M, Polascik TJ, Snyder DC, Ruffin MT, Moul JW, Brenner DE, Demark-Wahnefried W. Flaxseed-derived enterolactone is inversely associated with tumor cell proliferation in men with localized prostate cancer. J Med Food. 2013 Apr;16(4):357-60. doi: 10.1089/jmf.2012.0159. PMID 23566060
- [Result] Azrad M, Vollmer RT, Madden J, Polascik TJ, Snyder DC, Ruffin MT 4th, Moul JW, Brenner D, He X, Demark-Wahnefried W. Disparate results between proliferation rates of surgically excised prostate tumors and an in vitro bioassay using sera from a positive randomized controlled trial. Biotech Histochem. 2015 Apr;90(3):184-9. doi: 10.3109/10520295.2014.976840. Epub 2014 Dec 1. PMID 25434394